CLINICAL TRIAL: NCT05575245
Title: Clinical Of Drug-eluting Stent Versus Excimer Laser Ablation Combined Drug-coated Balloon To Treat Arteriosclerosis Occlusive Disease Of Lower Extremity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The research fund has not yet arrived.
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuH135
Record Dates: First submitted 2022-08-10; First posted 2022-10-12 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Atherosclerosis; Ischemia
Keywords: drug-eluting stent; debulking; femoral artery; drug-coated balloon
MeSH Terms: conditions — Atherosclerosis; Ischemia | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Drug-eluting Stent (Active Comparator): Drug-eluting Stent group
  Interventions: Device: Drug-eluting Stent
- Intervention: Excimer Laser Ablation Combined Drug-coated Balloon (Experimental): Excimer Laser Ablation Combined Drug-coated Balloon group
  Interventions: Device: Excimer Laser Ablation Combined Drug-coated Balloon

INTERVENTIONS:
Device: Drug-eluting Stent — Drug-eluting Stent angioplasty
  Arms: Intervention: Drug-eluting Stent
Device: Excimer Laser Ablation Combined Drug-coated Balloon — Excimer Laser Ablation Combined Drug-coated Balloon angioplasty
  Arms: Intervention: Excimer Laser Ablation Combined Drug-coated Balloon

SUMMARY:
This is a Prospective randomized controlled study to evaluate the difference of safety，effectiveness between Excimer Laser Ablation Combined Drug-coated Balloon and drug-eluting stent in treatment of femoral-popliteal artery lesions.

DETAILED DESCRIPTION:
Prospective randomized controlled study to evaluate the difference of safety，effectiveness between Excimer Laser Ablation Combined Drug-coated Balloon and drug-eluting stent in treatment of femoral-popliteal artery lesions. Patients with femoral-popliteal artery lesions in our department were randomly assigned to the Excimer Laser Ablation Combined Drug-coated Balloon group and drug-eluting stent group. Compare the ischemic improvement rate (limb salvage rate, postoperative patency rate) and the complications rate of two different treatments. At the same time, the peri-operative related factors that may affect the end point events, such as preoperative baseline data, lesion characteristics, imaging features, stent fracture, and end point observation indexes were analyzed by regression analysis.

ELIGIBILITY:
Inclusion criteria： 1.all patients signed an informed consent form; 2.digital subtraction angiography (DSA) revealed femoropopliteal artery stenosis above 70% or occlusion resulting in claudication (Rutherford clinical category-Becker class II-III2-3) or critical limb ischemia (CLI) (Rutherford clinical category 4-5-Becker class IV-V) 3.with unobstructed vascular inflow; 4.with at least a vessel runoff; 5. good compliance and regular follow-up.

Exclusion criteria: 1. Acute or subacute lower limb ischemia caused by acute intraluminal thrombus within the target lesion.; 2. Severe calcified lesions （grade 4 in the PACSS scale）; 3. In-stent restenosis lesion or surgical arterial bypass grafting; 4. Severe renal insufficiency: creatinine level greater than 2.5 mg/dL; 5. Platelet count below 100,000/μL or with antiplatelet / anticoagulation contraindications; 6. Immunologic diseases or malignant diseases; 7. Ongoing active infection; 8. Decompensated congestive heart failure or acute coronary syndrome; 9. Refuse to sign the informed consent Unwillingness to comply with follow-up suggestions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
12-month Primary Patency Rate | 12 months
  systolic velocity ratio >2.4 as measured by Duplex ultrasound.

SECONDARY OUTCOMES:
Technical success | 1 day
  Technical success was defined as residual stenosis less than 30% by final
freedom from clinically-driven TLR | 1 day
  it is defined as the freedom from clinically-driven target lesion revascularization
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation,
12-month Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China